CLINICAL TRIAL: NCT02228252
Title: Whey Protein, Postprandial Lipemia and Cardiovascular Disease: Evaluation of the Effect of a Pre-meal of Whey Protein on Postprandial Lipiemia in Subjects With the Metabolic Syndrome and Type 2 Diabetes
Brief Title: The Effect of Protein Quality and Time-factor by Consumption of a Pre-meal on Postprandial Lipemia in Subjects With the Metabolic Syndrome.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aarhus University Hospital (Other)
Collaborators: University of Aarhus (Other); University of Copenhagen (Other)
Responsible Party: Principal Investigator, Ann Bjørnshave, PhD student, Aarhus University Hospital
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: CERN-Premeal2
Record Dates: First submitted 2014-08-27; First posted 2014-08-28 (Estimated); Last update posted 2015-05-05 (Estimated); Status verified 2014-08

CONDITIONS: Metabolic Syndrome
Keywords: Proteins; Postprandial lipemia; Pre-meal; Metabolic syndrome
MeSH Terms: conditions — Metabolic Syndrome | interventions — Whey Proteins; Caseins; Glutens

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 20 g whey protein (-15 min) (Experimental): 20 g whey protein dissolved in 200 milliliter (mL) Water. Consumed as a pre-meal 15 min prior to the main meal.
  Interventions: Other: Whey protein
- 20 g whey protein (-30 min) (Experimental): 20 g whey protein dissolved in 200 milliliter (mL) Water. Consumed as a pre-meal 30 min prior to the main meal.
  Interventions: Other: Whey protein
- 20 g casein (Experimental): 20 g casein dissolved in 200 milliliter (mL) Water. Consumed as a pre-meal 15 min prior to the main meal.
  Interventions: Other: Casein
- 20 g gluten protein (Experimental): 21.5 g gluten protein dissolved in 200 milliliter (mL) Water. Consumed as a pre-meal 15 min prior to the main meal.
  Interventions: Other: Gluten protein

INTERVENTIONS:
Other: Whey protein
  Other Names: Brand name: LACPRODAN® SP-9225 Instant; Lot nr.: D150214
  Arms: 20 g whey protein (-15 min); 20 g whey protein (-30 min)
Other: Casein
  Other Names: Brand name: MIPRODAN 30; Lot nr.: 1594303
  Arms: 20 g casein
Other: Gluten protein
  Other Names: Brand name: Reppe wheat gluten
  Arms: 20 g gluten protein

SUMMARY:
Cardiovascular disease (CVD) is one of the most important and frequent causes of death. Postprandial lipidemia (PPL) is an independent risk factor for CVD, besides the traditional risk factors e.g. hypertension, high LDL-cholesterol, family disposition of CVD and type 2 diabetes (T2D). A high PPL is associated with an increased risk of myocardial infarction and stroke. Reduction of increased PPL, as a part of CVD prevention, is therefore pivotal. Especially in groups with increased risk of CVD, like the metabolic syndrome (MeS) and T2D. Identification of a simple diet-related method will possibly result in reduction of CVD in healthy as well as high-risk subjects.

The aim of this project is to investigate the effect of protein quality and the time factor of protein consumed as pre-meal prior to a fat-rich meal on responses of triglycerides and apolipoprotein B48 (ApoB48). Secondarily the aim is to study the responses of glucose, insulin, glucagon, amino acids, inflammatory markers, incretins, rate of gastric emptying and metabolomics. Also satiety feeling will be measured.

Investigators hypothesize that whey protein consumed 15 minutes prior to a fat-rich isocaloric meal reduces triglyceride- and ApoB48 responses more compared to casein protein and gluten protein consumed 15 minutes prior to the meal and whey protein consumed 30 minutes prior to the meal in subjects with MeS.

The investigators research will hopefully contribute to a better understanding of how PPL can be modified in a simple manner. It will promote innovation to the food industry for development and production of healthy food products, which can be applied in the fight against CVD in the background population in general and high-risk people in particular. Thus, the results of this project can impart knowledge of great importance both to the national and international food industry as well as the healthcare systems.

DETAILED DESCRIPTION:
Using a randomised, cross-over design 20 subjects with MeS will consume a test meal prior to a fat-rich meal. The test meals contain three different amounts of whey protein. Blood samples are collected before consumption of the pre-meal and after consumption of the fat-rich isocaloric meal during 360 minutes. The fat-rich isocaloric meal is a breakfast containing 1043 kcal (15 E% protein, 65 E% fat and 20 E% carbohydrates). The main-meal is composed of white bread, rye bread, butter, cheese (45 %), salami, egg, bacon, milk (1.5 % fat) and coffee (decaffeinated) and should be consumed over 15 min. Visual Analog Scale (VAS) will be used for determination of subjective satiety feeling.

ELIGIBILITY:
Inclusion Criteria:

- Central obesity (female > 80 cm; male > 94 cm) with two of the following parameters:

* Fasting triglycerides > 1.7 mmol/L
* Fasting HDL-cholesterol < 1.03 mmol/L (female) or <1.29 mmol/L (male)
* Blood pressure ≥ 130/85 mmHg
* Fasting plasma glucose ≥ 5.6 mmol/L Subjects who are in medical treatment with lipid and/or blood pressure-lowering habitual treatment can participate provided that the treatment is stable throughout the trial.

Exclusion Criteria:

* Type 1 diabetes
* Type 2 diabetes (HbA1c ≥ 48 mmol/L)
* Fasting plasma triglycerides > 5.0 mmol/L
* Blood pressure > 160/100 mmHg
* Cardiovascular, liver, kidney or metabolic disease
* Corticosteroid treatment
* Pregnancy or lactation
* Alcohol or drug abuse
* Legal incapacity

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2014-08; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Effect on triglyceride response of whey protein as pre-meal after a high-fat meal in subjects with the metabolic syndrome measured as incremental Area Under the Curve (iAUC -15 - 360 min). | Prior to the pre meal (-30/-15 min), prior to the main meal (0 min) and 60, 90, 120, 180, 240 and 360 min post main meal.
Effect on apolipoprotein B48 of whey protein as pre-meal after a high-fat meal in subjects with the metabolic syndrome measured as incremental Area Under the Curve (iAUC -15 - 360 min). | Prior to the pre meal (-30/-15 min), prior to the main meal (0 min) and 120, 240 and 360 min post main meal.

SECONDARY OUTCOMES:
Glucose responses measured as incremental Area Under the Curve (AUC -30/-15 - 360 min) | Prior to the pre meal (-30, -25) -15 min, (-10 min), prior to the main meal (0 min) and 15, 30, 60, 90, 120, 240 and 360 min post main meal.
Insulin responses measured as incremental Area Under the Curve (AUC -30/-15 - 360 min) | Prior to the pre meal (-30, -25) -15 min, (-10 min), prior to the main meal (0 min) and 15, 30, 60, 90, 120, 240 and 360 min post main meal.
Glucagon responses measured as incremental Area Under the Curve (AUC -30/-15 - 360 min) | Prior to the pre meal (-30, -25) -15 min, (-10 min), prior to the main meal (0 min) and 15, 30, 60, 90, 120, 240 and 360 min post main meal.
Glucagon-like peptide 1 (GLP-1) responses measured as incremental Area Under the Curve (AUC -30/-15 - 360 min) | Prior to the pre meal (-30, -25) -15 min, (-10 min), prior to the main meal (0 min) and 15, 30, 60, 90, 120, 240 and 360 min post main meal.
Gastric inhibitory peptide (GIP) responses measured as incremental Area Under the Curve (AUC -30/-15 - 360 min) | Prior to the pre meal (-30, -25) -15 min, (-10 min), prior to the main meal (0 min) and 15, 30, 60, 90, 120, 240 and 360 min post main meal.

OTHER OUTCOMES:
Responses of the inflammatory marker monocyte chemotactic protein-1 (MCP-1) measured as incremental Area Under the Curve (AUC -30/-15 - 360 min) | Prior to the pre meal (-30, -25) -15 min, (-10 min), prior to the main meal (0 min) and 15, 30, 60, 90, 120, 240 and 360 min post main meal.
Change in amino acids concentration from baseline to 30 min | Baseline (-30/-15 min), 30 min
Responses of free fatty acids measured as incremental Area Under the Curve (iAUC -30-15 - 360 min) | Prior to the pre meal (-30, -25) -15 min, (-10 min), prior to the main meal (0 min) and 15, 30, 60, 90, 120, 240 and 360 min post main meal.
Satiety measured as incremental Area Under the Curve (AUC -30/-15 - 360 min) | Prior to the pre meal (-30, -25) -15 min, (-10 min), prior to the main meal (0 min) and 15, 30, 60, 90, 120, 240 and 360 min post main meal.
  S-paracetamol
Responses of the inflammatory marker Rantes measured as incremental Area Under the Curve (AUC -30/-15 - 360 min) | Prior to the pre meal (-30, -25) -15 min, (-10 min), prior to the main meal (0 min) and 15, 30, 60, 90, 120, 240 and 360 min post main meal.
Responses of metabolomics measured as incremental Area Under the Curve (AUC -30/-15 - 360 min) in plasma. | Prior to the pre meal (-30/-15 min), prior to the main meal (0 min) and 120, 240 and 360 min post main meal.
Responses of metabolomics measured as incremental Area Under the Curve (AUC -30/-15 - 360 min) in urine. | Prior to the pre meal (-30/-15 min), and 120 and 360 min post main meal.
Responses of satiety visual analog scale (VAS) measured as incremental Area Under the Curve (AUC -30/-15 - 360 min) | Prior to the pre meal (-30/-15 min), prior to the main meal (0 min) and 30, 60, 90, 120, 150, 180, 210, 240, 270, 300 and 360 min post main meal

CONTACTS AND LOCATIONS:
Overall Officials: Kjeld Hermansen, Prefessor, Principal Investigator — Aarhus University Hospital
Locations (1):
- Aarhus University Hospital, Aarhus, Aarhus C, Denmark